CLINICAL TRIAL: NCT05522062
Title: Epidemiological Study for Traumatic Humeral Shaft Fractures in Adults Who Were Admitted to Assiut University Hospital Within One Year
Brief Title: Epidemiological Study for Traumatic Humeral Shaft Fractures in Adults
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Youssef Sameh, Principal Investigator, Assiut University
Other Study IDs: Humeral shaft fracture
Record Dates: First submitted 2022-08-27; First posted 2022-08-30 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Humerus Shaft Fracture
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgical treatment for humerus shaft fracture — surgical treatment for humerus shaft fracture

SUMMARY:
Primary Objective :

To evaluate the incidence of radial nerve palsy for adult patients with humeral shaft fractures

Secondary Objective :

To establish management protocol for traumatic humeral shaft fractures in adults at AUH

DETAILED DESCRIPTION:
Diaphyseal humeral shaft fracture is defined as an extra articular fracture of the humerus with Exclusion of both 5 cm of both upper and lower ends (Muller et al,1990) Within the last Century, many conservative and surgical techniques developed all over the world to solve this problem (Welter D et al, 1991) Conservative treatment was a gold standard since the full research which was published by Sarmiento (Sarmiento, 1977 ) Within the last few decades, with the establishment of osteosynthesis and surgical fixation of long bone which had better outcome in comparison to conservative treatment, it led to a changes in the protocols of treating fractures of the humerus (Muller et al,1990) Within the last decade, with the revolution of biological non anatomical fixation of the humeral shaft fractures, a new era of management was established and became popular all over the highly qualified trauma centres (Balam KM et al, 2014) So, the rational of this work, is to document different surgical strategies of biological fixation of humeral shaft fractures in adults with its results.

ELIGIBILITY:
Inclusion Criteria:

* All patients with traumatic humeral shaft fracture more than 16 years old who are admitted in Assiut University Hospital

Exclusion Criteria:

* Patients with humeral shaft fracture less than 16 years old or patients with pathological humeral shaft fracture

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Total coverage of all cases with inculsion criteria admitted to AUH in one year
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the occurrence of different patho-anatomic subtypes of humeral shaft fractures and the prevalence of primary radial nerve palsy clinically in patients preoperative and postoperative . | within one year
  To evaluate the occurrence of different patho-anatomic subtypes of humeral shaft fractures and the prevalence of primary radial nerve palsy clinically in patients preoperative and postoperative .

SECONDARY OUTCOMES:
To evaluate the effectiveness of surgical management for the different subtypes by follow up patients postoperative . | within one year
  To evaluate the effectiveness of surgical manag ement for the different subtypes by follow up patients postoperative .

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt

REFERENCES:
- [Background] Balam KM, Zahrany AS. Posterior percutaneous plating of the humerus. Eur J Orthop Surg Traumatol. 2014 Jul;24(5):763-8. doi: 10.1007/s00590-013-1355-2. Epub 2013 Nov 16. PMID 24241215
- [Background] Sarmiento A, Kinman PB, Galvin EG, Schmitt RH, Phillips JG. Functional bracing of fractures of the shaft of the humerus. J Bone Joint Surg Am. 1977 Jul;59(5):596-601. PMID 873955
- [Background] Updegrove GF, Mourad W, Abboud JA. Humeral shaft fractures. J Shoulder Elbow Surg. 2018 Apr;27(4):e87-e97. doi: 10.1016/j.jse.2017.10.028. Epub 2017 Dec 29. PMID 29292035
- [Background] Robinson CM, Hill RM, Jacobs N, Dall G, Court-Brown CM. Adult distal humeral metaphyseal fractures: epidemiology and results of treatment. J Orthop Trauma. 2003 Jan;17(1):38-47. doi: 10.1097/00005131-200301000-00006. PMID 12499966
- [Background] Horak J, Nilsson BE. Epidemiology of fracture of the upper end of the humerus. Clin Orthop Relat Res. 1975 Oct;(112):250-3. PMID 1192641